CLINICAL TRIAL: NCT00091234
Title: Gemtuzumab Ozogamicin (GO) Monotherapy Versus Standard Supportive Care for Previously Untreated AML in Elderly Patients Who Are Not Eligible for Intensive Chemotherapy: A Randomized Phase II/III Trial (AML-19) of the EORTC-LG and GIMEMA-ALWP
Brief Title: Gemtuzumab Ozogamicin in Treating Older Patients With Previously Untreated Acute Myeloid Leukemia
Acronym: AML-19
Status: Unknown | Phase: Phase 2 / Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: European Organisation for Research and Treatment of Cancer - EORTC (Network)
Collaborators: Gruppo Italiano Malattie EMatologiche dell'Adulto (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: EORTC-06031; EORTC-06031
Record Dates: First submitted 2004-09-07; First posted 2004-09-09 (Estimated); Last update posted 2012-07-24 (Estimated); Status verified 2012-07

CONDITIONS: Leukemia
Keywords: adult acute myeloid leukemia with 11q23 (MLL) abnormalities; adult acute myeloid leukemia with inv(16)(p13;q22); adult acute myeloid leukemia with t(16;16)(p13;q22); adult acute myeloid leukemia with t(8;21)(q22;q22); untreated adult acute myeloid leukemia; secondary acute myeloid leukemia; adult acute basophilic leukemia; adult acute eosinophilic leukemia; adult erythroleukemia (M6a); adult pure erythroid leukemia (M6b); adult acute megakaryoblastic leukemia (M7); adult acute minimally differentiated myeloid leukemia (M0); adult acute monoblastic leukemia (M5a); adult acute monocytic leukemia (M5b); adult acute myeloblastic leukemia with maturation (M2); adult acute myeloblastic leukemia without maturation (M1); adult acute myelomonocytic leukemia (M4)
MeSH Terms: conditions — Leukemia; Congenital Abnormalities; Leukemia, Basophilic, Acute; Leukemia, Eosinophilic, Acute; Leukemia, Erythroblastic, Acute; Leukemia, Megakaryoblastic, Acute; Leukemia, Monocytic, Acute; Leukemia, Myeloid, Acute; Leukemia, Myelomonocytic, Acute | interventions — Gemtuzumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Drug: gemtuzumab ozogamicin

SUMMARY:
RATIONALE: Monoclonal antibodies such as gemtuzumab ozogamicin can locate cancer cells and either kill them or deliver cancer-killing substances to them without harming normal cells. It is not yet known whether gemtuzumab ozogamicin is more effective than standard supportive care in treating older patients who have acute myeloid leukemia.

PURPOSE: This randomized phase II/III trial is studying two different gemtuzumab ozogamicin regimens to see how well they work compared to standard supportive care in treating older patients with previously untreated acute myeloid leukemia.

DETAILED DESCRIPTION:
OBJECTIVES:

* Compare the feasibility, toxicity, and antileukemic activity of two different dosing regimens of gemtuzumab ozogamicin (GO) vs standard supportive care in older patients with previously untreated acute myeloid leukemia who are not candidates for intensive chemotherapy. (phase II)
* Compare the efficacy and toxicity of the best dosing regimen of GO selected from phase II vs standard supportive care, in terms of overall survival, in these patients. (phase III)

OUTLINE: This is a randomized, open-label, multicenter phase II study followed by a phase III study. Patients are stratified according to age (61 to 75 vs 76 to 80 vs 81 and over), CD33-positivity of bone marrow blasts (< 20% vs 20-80% vs > 80% vs unknown), initial WBC before hydroxyurea administration (< 30,000/mm^3 vs ≥ 30,000/mm^3), WHO performance status (0-1 vs 2 vs 3-4), and participating center.

* Phase II: Patients are randomized to 1 of 3 treatment arms.

  * Arm I: Patients receive gemtuzumab ozogamicin (GO) IV over 2 hours on days 1 and 8. Patients with stable or responding disease at day 36 receive GO IV over 2 hours every 4 weeks for up to 8 courses in the absence of disease progression or unacceptable toxicity.
  * Arm II: Patients receive GO IV over 2 hours on days 1, 3, and 5. Patients with stable or responding disease at day 36 receive GO IV over 2 hours every 4 weeks for up to 8 courses in the absence of disease progression or unacceptable toxicity.
  * Arm III: Patients receive standard supportive care.
* Phase III: Patients are randomized to 1 of 2 treatment arms.

  * Arm I: Patients receive the selected treatment (arm I or arm II) from phase II.
  * Arm II: Patients receive standard supportive care. Patients who receive GO treatment are followed monthly for 1 year and then every 3 months thereafter. Patients who receive standard supportive care are followed at least every 4 weeks.

PROJECTED ACCRUAL: A total of 259 patients (75 for phase II [25 per treatment arm] and 184 for phase III [92 per treatment arm]) will be accrued for this study within 2.5 years.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically confirmed acute myeloid leukemia (AML)

  * At least 20% bone marrow blasts by bone marrow aspiration or biopsy
  * All subtypes except M3 (acute promyelocytic leukemia) are allowed
* Previously untreated primary or secondary disease (including AML after myelodysplastic syndromes)
* Ineligible for intensive chemotherapy, as defined by 1 of the following criteria:

  * 61 to 75 years old AND WHO performance status > 2 AND/OR unwilling to receive intensive chemotherapy
  * Over 75 years old
* No blast crisis of chronic myeloid leukemia
* No AML supervention after other myeloproliferative disease
* WBC < 30,000/mm^3 and meets 1 of the following criteria:

  * WBC < 30,000/mm^3 at diagnosis AND had no prior treatment with hydroxyurea
  * WBC ≥ 30,000/mm^3 at diagnosis AND received mandatory pretreatment with hydroxyurea (up to 14 days duration) until WBC < 30,000/mm^3
* No active CNS leukemia

PATIENT CHARACTERISTICS:

Age

* See Disease Characteristics
* 61 and over

Performance status

* See Disease Characteristics

Life expectancy

* Not specified

Hematopoietic

* See Disease Characteristics

Hepatic

* Bilirubin ≤ 1.5 times upper limit of normal (ULN)

Renal

* Creatinine ≤ 1.5 times ULN

Cardiovascular

* No arrhythmia requiring chronic treatment
* No congestive heart failure
* No symptomatic ischemic heart disease
* No other severe cardiovascular disease

Pulmonary

* No severe pulmonary dysfunction ≥ grade 3

Other

* No alcohol abuse
* No severe neurological or psychiatric disease
* No active uncontrolled infection or severe systemic infection
* No other malignancy
* No psychological, familial, sociological, or geographical condition that would preclude study compliance and follow-up
* HIV negative

PRIOR CONCURRENT THERAPY:

Biologic therapy

* No concurrent filgrastim (G-CSF) or sargramostim (GM-CSF)
* No concurrent antiangiogenic drugs

Chemotherapy

* See Disease Characteristics
* Concurrent low-dose cytostatic agents (i.e., thioguanine or mercaptopurine) allowed for palliative care (standard supportive care arm only)

Endocrine therapy

* Prior corticosteroids (duration ≤ 14 days ) for primary or secondary AML allowed

Radiotherapy

* Not specified

Surgery

* Not specified

Other

* No other concurrent cytotoxic drugs
* No other concurrent experimental therapy
* No concurrent tyrosine kinase inhibitors

Min Age: 61 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 279 (Estimated)
Dates: Start 2004-06; Primary Completion 2013-12 (Estimated)

PRIMARY OUTCOMES:
Proportion of patients able to start continuation therapy (Phase II)
Overall survival (Phase III)

SECONDARY OUTCOMES:
Rate of complete remission (CR+CRp)by the end of continuation therapy, for patients in the GO arms (Phase II)
Overall survival (Phase II)
Toxicity (CTCAE grading), including time to hematological recovery (Phase II & III)
Rate of complete remisison (CR+CRp) by the end of induction and by the end of continuation therapy, for patients in GO arm (Phase III)
Disease-free survival for patients who reached CR or CRp (Phase III)
Progression-free survival from randomization for patients in GO arm (Phase III)

CONTACTS AND LOCATIONS:
Overall Officials: Sergio Amadori, MD, Principal Investigator — EORTC - AZIENDA OSPEDALLERA UNIVERSITARIA - POLICLINICO TOR VERGATA, IT; Giuliana Alimena, Principal Investigator — GIMEMA - Universita Degli Studi "La Sapeinza"
Locations (45):
- Belgium (7):
  - Ziekenhuis Netwerk Antwerpen Middelheim, Antwerp
  - AZ Sint-Jan, Bruges
  - Institut Jules Bordet, Brussels
  - Hopital Universitaire Erasme, Brussels
  - Universitair Ziekenhuis Antwerpen, Edegem
  - CHU Liege - Domaine Universitaire du Sart Tilman, Liège
  - Centre Hospitalier Peltzer-La Tourelle, Verviers
- Italy (34):
  - Ospedale S Donato, USL-8, Arezzo Cap
  - Universita Degli Studi di Bari, Bari
  - Universita Di Brescia, Brescia
  - Ospedale Binaghi, Cagliari
  - Ospedale Oncologico A. Businco, Cagliari
  - Ospedale Regionale A Pugliese, Cantanzaro
  - Ospedale Ferrarotto, Catania
  - Ospedale Regionale A. Pugliese, Catanzaro
  - Universita di Ferrara, Ferrara
  - Azienda Ospedaliera Vito Fazzi, Lecce
  - Azienda Ospedaliera - Universitaria di Modena, Modena
  - Ospedale Di Montefiascone, Montefiascone
  - Azienda Ospedaliera di Rilievo Nazionale A.Cardarelli, Naples
  - Ospedale Maggiore della Carita, Novara
  - Azienda Ospedaliera Policlinico Paolo Giaccone, Palermo
  - Ospedale La Maddalena - Palermo, Palermo
  - Azienda Ospedaliera Di Parma, Parma
  - Policlinico Monteluce, Perugia
  - Ospedale San Salvatore, Pesaro
  - Ospedale Civile Pescara, Pescara
  - Ospedale San Carlo, Potenza
  - Ospedale Sta. Maria Delle Croci, Ravenna
  - Ospedale Sant'Andrea, Roma
  - Azienda Ospedaliera Universitaria Policlinico Tor Vergata, Rome
  - Ospedale Sant' Eugenio, Rome
  - Libero Istituto Universitario Campus Bio-Medico, Rome
  - Azienda Policlinico Umberto Primo, Rome
  - Istituto Regina Elena, Rome
  - Policlinico A. Gemelli - Universita Cattolica del Sacro Cuore, Rome
  - H. San Giovanni-Addolorata Hospital, Rome
  - Universita Degli Studi "La Sapeinza", Rome
  - Istituto di Ematologia Universita - University di Sassari, Sassari
  - Universita di Siena, Siena
  - Ospedale Maggiore dell' Universita, Trieste
- Netherlands (4):
  - Jeroen Bosch Ziekenhuis, 's-Hertogenbosch
  - Onze Lieve Vrouwe Gasthuis, Amsterdam
  - Leiden University Medical Center, Leiden
  - Universitair Medisch Centrum St. Radboud - Nijmegen, Nijmegen

REFERENCES:
- [Result] Amadori S, Suciu S, Selleslag D, et al.: Phase II-III study of gemtuzumab ozogamicin monotherapy versus best supportive care in older patients with newly diagnosed AML unfit for intensive chemotherapy: first results of the EORTC-GIMEMA AML-19 trial. [Abstract] Blood 112 (11): A-762, 2008.
- [Derived] Amadori S, Suciu S, Selleslag D, Aversa F, Gaidano G, Musso M, Annino L, Venditti A, Voso MT, Mazzone C, Magro D, De Fabritiis P, Muus P, Alimena G, Mancini M, Hagemeijer A, Paoloni F, Vignetti M, Fazi P, Meert L, Ramadan SM, Willemze R, de Witte T, Baron F. Gemtuzumab Ozogamicin Versus Best Supportive Care in Older Patients With Newly Diagnosed Acute Myeloid Leukemia Unsuitable for Intensive Chemotherapy: Results of the Randomized Phase III EORTC-GIMEMA AML-19 Trial. J Clin Oncol. 2016 Mar 20;34(9):972-9. doi: 10.1200/JCO.2015.64.0060. Epub 2016 Jan 25. PMID 26811524